CLINICAL TRIAL: NCT04513626
Title: A Randomized Comparative Phase II Trial Evaluating the Capacity of the Dual Combination Doravirine/Raltegravir to Maintain Virological Success in HIV-1 Infected Patients With an HIV-RNA Plasma Viremia Below 50 Copies/mL Under a Current Antiretroviral Regimen
Brief Title: HIV-1 Infected Patients, Phase II Trial, Dual Combination Doravirine/Raltegravir Open Label
Acronym: DORAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 010
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — doravirine; Raltegravir Potassium

STUDY DESIGN:
Intervention Model Description: This study is an open label, randomized, switch study, over 96 weeks, in which virally suppressed patients on a stable combined ART regimen will be randomized (2:1) to an immediate switch to doravirine/raltegravir (immediate switch group) or to the maintaining of their current ART followed by a switch to doravirine/raltegravir at W48 (delayed switch group). Patients will be followed during 96 weeks.
  The randomization will be stratified on gender and antiretroviral regimen at inclusion (Dual therapy or more).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed switch (Other): the maintaining of their current ART followed by a switch to doravirine/raltegravir at W48 (delayed switch group).
  Interventions: Drug: DORAVIRINE 100 MG [Pifeltro]
- Immediate switch (Experimental): Immediate switch to doravirine/raltegravir
  Interventions: Drug: DORAVIRINE 100 MG [Pifeltro]

INTERVENTIONS:
Drug: DORAVIRINE 100 MG [Pifeltro] — Immediate switch
  Other Names: Raltegravir 600 Mg x 2 [Isentress]

SUMMARY:
The objective of antiretroviral therapy (ART) is the maintenance of HIV viral suppression, the optimal condition to prevent disease progression, to optimize immune restoration, to prevent the development of viral resistance and to reduce viral transmission. Antiretroviral therapy has to be maintained long life over decades in the absence of strategies for HIV cure. This is why the long-term cumulative toxicity of ARV drugs is a major issue. Indeed as a consequence of potent ART strategies, in 2011 over 88% of patients on ART in the French Hospital database (ANRS CO4 FHDH) achieved viral suppression with HIV-RNA plasma viral load < 50 copies/mL and nearly 60% had CD4 > 500/mm3. As a consequence of massive reduction of mortality and morbidity related to HIV, infected patients are aging with 40% of patients over 50 years of age in the ANRS CO4 FHDH.

The current standard-of-care for antiretroviral therapy consists in a triple drug combination with two nucleoside reverse transcriptase inhibitors (NRTIs) plus either a non-nucleoside reverse transcriptase inhibitor (NNRTI), a protease inhibitor (PI), or an integrase inhibitor (INSTI). NRTIs and PIs have been associated to cumulative long-term toxicity such as bone and renal disorders related to tenofovir and increased cardio-vascular risk with PIs. In general population, aging is associated with well-known comorbidities such as bone demineralization, increased incidence of cardio or cerebrovascular disease, diabetes, renal dysfunction. HIV infected patients are at a greater risk for such abnormalities. Another crucial concern is the high probability of drug-drug interactions in HIV-infected patients, between ART and comedications.

Alternative strategies are needed, which must address the following questions: how to maintain the control of HIV viral replication while minimizing the occurrence of long-term clinical and metabolic complications, and minimizing the risk of drug-drug interactions?

This study is an open label, randomized, switch study over 96 weeks in which virally suppressed patients on a stable combined ART regimen will be randomized (2:1) to an immediate switch to doravirine/raltegravir (immediate switch group) or to the maintaining of their current ART followed by a switch to doravirine/raltegravir at W48 (delayed switch group). Patients will be followed during 96 weeks.

DETAILED DESCRIPTION:
The recent years have highlighted the cumulative toxicities of long-term exposure to antiretroviral drugs. Cardiovascular disease is one of the most common comorbidities in the aging HIV-infected population. Coronary artery disease (CAD) results from a combination of increasing age, traditional risk factor such as smoking, toxicity from long-term ART, and potentially related to HIV immune activation.

Most of boosted PIs and the NNRTI [efavirenz] are associated to an increase in triglycerides and total cholesterol plasma levels. In the ANRS CO8 APROCO COPILOTE cohort about 30% of patients developed hypertriglyceridemia. Prevalence of lipodystrophy and metabolic alterations and these alterations appear as early as 12 months after the initiation of PI therapy.

The prevalence of osteopenia and osteoporosis in HIV-infected individuals is higher in HIV-infected compared with HIV-negative individuals ranging, from 23 to 65% for osteopenia and from 3 to 22% for osteoporosis according to the studies [13-16] with, as consequence, a higher prevalence of patients with fracture (p < 0.0001).

Tenofovir is currently the most widely used antiretroviral drug. Globally, clinical trials have suggested that renal toxicity related to tenofovir is low (approximately 1%) in selected populations from clinical studies. However, observational cohort studies have suggested that this risk was higher with rates varying from approximately 2%.

In a systematic review and meta-analysis whereas over time with longer exposure to antiretroviral drugs the overall relative risk of renal disease was 3.87 (95% CI: 2.85-6.85) in HIV-infected patients compared to HIV-uninfected in ART treated patients. 0.54 (95% CI: 0.29-0.99) compared to naïve patients and 1.56 (95% CI: 0.83-2.93) in patients treated with tenofovir compared to patients without tenofovir.

In the DAD study not only tenofovir but also abacavir, lopinavir/ritonavir and atazanavir/ritonavir were associated to high risk.

The use of strategies that could minimize renal toxicity has to be investigated particularly in senior HIV infected population.

Increased risk for drug-drug interactions: a cause of concern in the elderly. Aging increases polypharmacy prescriptions for treatment and prevention of comorbidities such as cardio-vascular disease, hypertension or diabetes. One major issue is the risk for drug-drug interactions in elderly ART treated HIV infected patients due to the common CYP450 cytochrome pathway, shared by ARV drug and drug for comorbidities.

Monitoring concentration of these drugs is not easy in routine practice. Given these drug-drug interactions with potential severe clinical consequences, it is key to investigate alternative ART strategies with different metabolization pathways, such as raltegravir.

Raltegravir and Doravirine: benefits and advantages in terms of toxicity. Overall, literature data showed that raltegravir and doravirine are two drugs with high antiretroviral potency, including in experienced HIV-treated patients, with very good tolerance profile and without expected drug-drug interaction between the two drugs. A new dual therapy strategy combining doravirine + raltegravir given once daily has to be evaluated.

In the setting of dual therapies, and as background the excellent results in terms of efficacy of doravirine plus raltegravir (<2% of virological failure (95% confidence interval 0.3 to 5.0) at week 96 of 165 participants in the ETRAL), we postulate that:

* The association of raltegravir 1200 mg QD and doravirine 100 mg QD (DOR/RAL) will maintain viral suppression in HIV-1-infected patients with suppressed viremia on ART, with a virological failure rate of <12% in a population of 100 patients
* DOR/RAL will be associated to a robust viral suppression with limited amount of blips
* DOR/RAL will be well tolerated over the study period
* Acquired resistance to doravirine or raltegravir will be limited in case of virological failure
* DOR/RAL will present a benefit for patients on metabolic parameters and general symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with HIV-1 documented infection
* CD4 ≥ 200/mm3
* On stable combined ART regimen with at least 2 drugs for at least 6 months
* HIV-RNA plasma VL ≤ 50 copies/mL during the last 12 months prior to screening visit (W-6/W-4), documented by at least 2 time-points with no more than one blip (defined as one HIV-RNA plasma VL between 51 and 200 copies/mL followed by one HIV-RNA plasma VL ≤ 50 copies/mL)
* Naive to doravirine
* Absence of resistance to doravirine* and/or raltegravir**(see list mutations below)

  * on all HIV-genotypes with available RT and integrase gene sequences allowing resistance interpretation in case of previous virological failure
  * or on DNA genotype performed at screening if HIV genotype is not available in case of prior virological failure.
* Signed informed consent form.
* Patient affiliated to a social insurance regimen. For French patients only: subject enrolled in or a beneficiary of a Social Security programme (State Medical Aid or AME is not a Social Security programme).

  * Mutations associated to doravirine resistance are: V106A/M, Y188L, G190E/S, M230L, F227C, at least 2 among: A98G, L100I, K101E, V106I, E138K, Y181C/V, G190A or H221Y

    * Mutations associated to raltegravir resistance are: T66A/K, E92Q, G118R, F121Y, G140A/S Y143A/C/G/H/R/S, Q148E/G/H/K/R, V151L, N155H/S/T, E157Q, S230R, R263K, L74 F/I + V75I.

Exclusion Criteria:

* Absence of RT and INI HIV sequence available (past genotypes or failure of amplification of DNA at screening)
* HBV co-infection
* Hemoglobin <9 g/dL
* Platelets <80,000/mm3
* Creatinine clearance <60 mL/min (MDRD)
* AST or ALT ≥5N
* Concomitant DAA for anti-HCV therapy
* Any severe concomitant illness
* Any drug with potential drug-drug interaction with doravirine
* Concomitant treatment using interferon, interleukins or any other immune-therapy or chemotherapy
* Concomitant prophylactic or curative treatment for an opportunistic infection
* All conditions (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with trial protocol compliance, adherence and/or trial treatment tolerance
* Subjects under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship
* Subjects participating in another clinical trial evaluating different therapies and including an exclusion period that is still in force during the screening phase
* Pregnant women or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Measure the virological efficacy at week 48 of once daily doravirine plus raltegravir dual therapy to assess the effectiveness of the dual therapy DORAL to maintain the virological success to W48 | 48 weeks
  Measure of plasma viral load assessed by RNA quantification using COBA 6800 system (Roche)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Pitie-Salpetriere Hospital
Locations (1):
- Christine KATLAMA, Paris, Île-de-France Region, France